CLINICAL TRIAL: NCT04943315
Title: Clinical Evaluation of Monolithic Zirconia and Metal-ceramic Posterior Crowns
Brief Title: Clinical Evaluation of Monolithic Zirconia Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Kuraray Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University Complutense Madrid; 4157246 (Other Grant/Funding Number: Kuraray Europe GmbH)
Record Dates: First submitted 2021-06-23; First posted 2021-06-29 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Dental Materials
Keywords: crowns; metal-ceramic; monolithic zirconia; clinical evaluation; survival; wear
MeSH Terms: interventions — Metal Ceramic Alloys

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monolithic zirconia (Experimental): To assess the clinical performance and survival of posterior monolithic zirconia crowns
  Interventions: Procedure: Monolithic zirconia
- Metal-ceramic (Active Comparator): To assess the clinical performance and survival of posterior metal-ceramic crowns
  Interventions: Procedure: Metal-ceramic

INTERVENTIONS:
Procedure: Monolithic zirconia — posterior crowns
  Other Names: Katana
  Arms: Monolithic zirconia
Procedure: Metal-ceramic — posterior crowns
  Arms: Metal-ceramic

SUMMARY:
The objectives of the present study are to compare the survival rates and possible biological and technical complications of metal-ceramic, and monolithic third-generation zirconia posterior crowns. The null hypothesis is that no diﬀerences would be found between the parameters studied for each type of restoration.

DETAILED DESCRIPTION:
Seventy patients requiring at least one crown in the posterior region of the maxilla or mandible were included in this study. All subjects were recruited from the Master in Buccofacial Prostheses and Occlusion (Faculty of Odontology, University Complutense of Madrid, Spain). Before treatment, patients were informed of the study objectives, clinical procedures, materials used, advantages and possible risks of the ceramic material, and other therapeutic alternatives. Prior to the study, participants were asked to provide written informed consent. Seventy posterior crowns were produced and allocated in parallel and randomly to either monolithic third-generation zirconia, or metal-ceramic (MC) restorations. The clinical procedures were performed by two experienced clinicians. All participants received oral hygiene instructions and a professional tooth cleaning prior to prosthetic treatment. The abutment teeth were prepared with a 0.8- to 1-mm-wide circumferential chamfer, an axial reduction of 1 mm and an occlusal reduction of 1- to 2.0-mm. A 10- to 15- degree angle of convergence was achieved for the axial walls. Tooth preparations were scanned with an intraoral scanner and the crowns were designed using speciﬁc software. The restorations were then cemented using a resin self-adhesive cement. After cementation, occlusal contacts were evaluated, and the adjusted surfaces were polished using a porcelain polishing kit. The 70 crowns were examined at 1week (baseline),1, 2 and 3 years by 2 researchers who were not involved in the restorative treatment.

ELIGIBILITY:
Inclusion Criteria:

* One posterior tooth (molar or premolar) to be crowned
* Vital abutment or abutment with an adequate endodontic treatment
* Abutment not crowned previously
* Periodontally healthy abutment with no signs of bone resorption or periapical disease.
* Adequate occlusogingival height ≥ 4 mm.
* Stable occlusion and the presence of natural antagonist tooth.

Exclusion Criteria:

* Patients who present reduced crown length (less than 4 mm occlusogingival height).
* Poor oral hygiene, high caries activity, or active periodontal disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Quality of restorations at baseline | Baseline
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's (CDA) assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Quality of restorations at 1 year | 1 year
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's (CDA) assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Quality of restorations at 2 years | 2 years
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's (CDA) assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Quality of restorations at 3 years | 3 years
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's (CDA) assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Plaque Index (PI) at baseline | baseline
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 1 year | 1 year
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 2 years | 2 years
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 3 years | 3 years
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at baseline | Baseline
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 1 year | 1 year
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 2 years | 2 years
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 3 years | 3 years
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Margin stability at baseline | Baseline
  To assess the gingival margin stability throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 1 year | 1 year
  To assess the gingival margin stability throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 2 years | 2 years
  To assess the gingival margin stability throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 3 years | 3 years
  To assess the gingival margin stability throughout the evaluation period (subgingival, isogingival or supragingival)
Probing depth at baseline | Baseline
  Probing depth of the abutment and control teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 1 year | 1 year
  Probing depth of the abutment and control teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 2 years | 2 years
  Probing depth of the abutment and control teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 3 years | 3 years
  Probing depth of the abutment and control teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome
Patient satisfaction at 3 years | 3 years
  Subjective patient satisfaction using Visual analogue scale (VAS) ranged from 0 (worst possible result) to10 (best possible result). The items analyzed were: esthetics, function, comfort, overall satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Suarez, PhD, Study Director — Universidad Complutense de Madrid
Locations (1):
- Faculty of Odontology, Madrid, Spain